CLINICAL TRIAL: NCT01587482
Title: PacLitaxel Eluting Balloon Application In Sfa In Stent Restenosis
Acronym: PLAISIR
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROG/11/79
Record Dates: First submitted 2012-02-15; First posted 2012-04-30 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Peripheral Arterial Disease
Keywords: Superficial femoral artery; endovascular; Drug eluting balloon; Paclitaxel
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- drug eluting balloon: In this observationnal study, the intervention of interest is the use of drug eluting balloon in stent restenosis.
  Only the treated patients were included in this cohort.
  Interventions: Procedure: PacLitaxel Eluting Balloon Application

INTERVENTIONS:
Procedure: PacLitaxel Eluting Balloon Application — Stenting is a standard of care in revascularization for superficial femoral artery (SFA) atherosclerotic lesions. However, the Achilles' heel of this technique remains in-stent restenosis (ISR). While most of local therapies have failed to demonstrate significant benefit, studies for the treatment of SFA ISR are lacking and percutaneous transluminal angioplasty remains the current standard of care for this indication. Recent studies have shown successful results of drug eluting balloon in the treatment of SFA de-novo lesions and of coronary ISR.

SUMMARY:
Nowadays, stenting is became a standard of care in revascularization for superficial femoral artery (SFA) atherosclerotic lesions. However, the Achilles' heel of this technique remains in-stent restenosis (ISR). While most of local therapies have failed to demonstrate significant benefit, studies for the treatment of SFA ISR are lacking and percutaneous transluminal angioplasty remains the current standard of care for this indication. Recent studies have shown successful results of drug eluting balloon in the treatment of SFA de-novo lesions and of coronary ISR. FREERIDE, a French prospective cohort has been set up to evaluate the safety and the efficacy of drug eluting balloon (DEB) for the treatment of SFA atherosclerotic lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Symptomatic patient according to Rutherford Class 1, 2, 3, 4 or 5
* Clinical degradation by at least 1 Rutherford stage or absence of healing of all skin lesions
* Symptoms related to SFA ISR defined by PSVR > 2.4 within 3 to 24 months after SFA stenting of de novo atherosclerotic lesions. Each patient may have either one or both limbs treated in the study
* The target ISR lesion is fully comprised between the origin of the SFA and distally the femoropopliteal crossover (crossing by SFA of medial rim of femur in the PA projection)
* Adequate SFA inflow and outflow either pre-existing or successfully re-established (outflow defined as patency of at least one infragenicular artery)
* The target lesion must no extend beyond the stent margin
* Successful crossing of the target lesion, inflow and outflow lesions with a guidewire
* Patient belongs to the French health care system
* Written informed consent

Exclusion Criteria:

* No atheromatous disease
* Asymptomatic lesion
* Known allergies to heparin, aspirin, other anti-coagulant/antiplatelet therapies, and/or paclitaxel
* Acute limb ischemia
* Patient on oral anticoagulation therapy
* Target lesion requires / has been pre-treated with alternative therapy such as: DES, laser, atherectomy, cryoplasty, cutting/scoring balloon, etc.
* Life expectancy < 1 year
* Patient involved in another trial
* Refusing patient
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From December 2011 to December 2012 at 13 hospitals in France, we will include patients with symptomatic atherosclerotic lesions related to superficial femoral artery in-stent restenosis to undergo endovascular repair by paclitaxel drug eluting balloon. 100 patients will be included.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Target Lesion Revascularization (TLR) | at 1 year

SECONDARY OUTCOMES:
Major Adverse Events through | at 1 year
Target extremity revascularization (TER) | at 1, 3, 6, 9, 12 and 18 months after surgery
clinical improvement equal or above to a stage according to Rutherford classification without superficial femoral artery revascularization | at 1, 3, 6, 9, 12 and 18 months
  to assess primary maintenance of clinical improvement
peak systolic velocity index without Target Lesion Revascularization | at 1, 3, 6, 9, 12 and 18 months
  to assess primary patency
Quality of life assessment by EQ5D questionnaire | at 1, 3, 6, 9, 12 and 18 mois after surgery
post-angioplasty restenosis | at 1, 3, 6, 9, 12 and18 months after surgery
drug relief success without balloon break | during surgery
Length of hospitalization stay | at 1 year
clinical improvement equal or above to a stage according to Rutherford classification with possible superficial femoral artery surgery | at 1, 3, 6, 9, 12 and 18 months
  to assess secondary maintenance of clinical improvement
peak systolic velocity index | at 1 year
  to assess secondary patency
intra-stent restenosis | at 1, 3, 6, 9, 12 and 18 months after surgery
  significant whether restenosis >50% and peak systolic velocity index > 2.4

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Reix, PU-PH, Principal Investigator — Amiens's Univeristy Hospital; Eric Ducasse, PU-PH, Principal Investigator — Pellegrin's University Hospital; Patrick Lermusiaux, PU-PH, Principal Investigator — Lyon's University Hospital; Jean-Marc Pernes, Practitioner, Principal Investigator — Antony's private Hospital; Nicolas Louis, PH, Principal Investigator — Le Raincy-Montfermeuil Hospital; Antoine Sauget, Practitioner, Principal Investigator — Pasteur's private Hospital; Philippe Commeau, Practitioner, Principal Investigator — Ollioules private Hospital; Jean-Noel Albertini, PU-PH, Principal Investigator — St Etienne University Hospital; Olivier Planché, PH, Principal Investigator — Le Plessis-Robinson private hospital (CMC); Max Amor, PH, Principal Investigator — Essey-les-Nancy Private hospital (Polyclinique Pasteur); Jean-Marie Cardon, Dr, Principal Investigator — Nimes private Hospital (clinique des fransiscaines); Alain Cardon, PH, Principal Investigator — Rennes's University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Bague N, Julia P, Sauguet A, Pernes JM, Chatelard P, Garbe JF, Penillon S, Cardon JM, Commeau P, Planche O, Guyomarch B, Goueffic Y. Femoropopliteal In-stent Restenosis Repair: Midterm Outcomes After Paclitaxel Eluting Balloon Use (PLAISIR Trial). Eur J Vasc Endovasc Surg. 2017 Jan;53(1):106-113. doi: 10.1016/j.ejvs.2016.10.002. Epub 2016 Nov 24. PMID 27890526